CLINICAL TRIAL: NCT06811220
Title: The Effect of Oral Administration of Hesperidin and Diosmin in Reducing Paclitaxel-induced Peripheral Neuropathy in Breast Cancer Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0108808
Record Dates: First submitted 2025-01-28; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Paclitaxel-induced peripheral neuropathy
MeSH Terms: conditions — Breast Neoplasms | interventions — Diosmin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Control group): 70 patients will receive Paclitaxel only as neoadjuvant chemotherapy as one (No Intervention): Patients will receive Paclitaxel only as neoadjuvant chemotherapy as one cycle every 21 days (i.e. 3 weeks) as 175 mg/m2.
- Group 2 (Intervention group): patients which will receive Paclitaxel plus Hespiridin and Diosmin. (Active Comparator): patients which will receive Paclitaxel plus Daflon® (50 mg Hesperidin and Micronized purified flavonoid fraction (MPFF) 450 diosmin combination one film coated tablet) 2 tablets daily, i.e. 1 tablet at midday and 1 tablet in the evening, at meal times.
  Interventions: Drug: Hespiridin and Diosmin

INTERVENTIONS:
Drug: Hespiridin and Diosmin — Daflon® (50 mg Hesperidin and Micronized purified flavonoid fraction (MPFF) 450 diosmin combination one film coated tablet)
  Arms: Group 2 (Intervention group): patients which will receive Paclitaxel plus Hespiridin and Diosmin.

SUMMARY:
The aim of this study is evaluation of the potential neuroprotective effect of oral hesperidin and diosmin in reducing paclitaxel- induced peripheral neuropathy in the treatment of breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients over 18 years of age with pathologically confirmed breast cancer.
2. Breast cancer patients candidate for chemotherapy and will receive paclitaxel.
3. Patients having an eastern cooperative oncology group (ECOG) score more than 2

Exclusion Criteria:

1. Patients with signs and symptoms of clinical neuropathy at baseline.
2. Patients with diabetes mellitus, alcoholic disease, heart failure, pregnant or lactating women.
3. Patients receiving vitamin/ supplementation drugs that interfere with the study intervention.
4. Patients who have previously received chemotherapy.
5. Hepatic impaired patients.
6. Patient with history of allergy to hesperidin.
7. Patients with history of allergy to diosmin.
8. Renal impaired patients.
9. Patient inadherent to paclitaxel.
10. Patients inadherent to the administered hesperidin and diosmin during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patients
Enrollment: 140 (Estimated)
Dates: Start 2025-01-27 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in serum levels of the following biomarker:Nerve growth factor (NGF) | 3 months
  Nerve growth factor (NGF) measured in Pg/ml
Changes in serum levels of the following biomarker :Malondialdehyde (MDA). | 3 months
  Malondialdehyde (MDA) is measured in Micro mole/L
Changes in serum levels of the following biomarker:Interleukin-1 beta (IL-1 β). | 3 months
  Interleukin-1 beta (IL-1 β) is measured in Pg/ml
Changes in serum levels of the following biomarker: Tumor necrosis Factor-Alpha (TNF- α) . | 3 months
  Tumor necrosis Factor-Alpha (TNF- α) is measured in Pg/ml

SECONDARY OUTCOMES:
A- Incidence of chemotherapy induced-peripheral neuropathy using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria assessed. | at baseline and after each cycle of neoadjuvant chemotherapy where the length of each cycle is 21 days (i.e. every 21 days).
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria ; where its classified as mild, moderate and severe peripheral neuropathy according to severity of subjective peripheral neuropathy reported by the patient.
B- Measurement of the quality of life using the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity FACT/GOG-NTX (Version 4) questionnaire assessed. | at baseline and after each cycle of neoadjuvant chemotherapy where the length of each cycle is 21 days (i.e. every 21 days).
  Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity FACT/GOG-NTX (Version 4) questionnaire where the minumum score is zero and the maximum score is 16. The higher the score the better the quality of life.